CLINICAL TRIAL: NCT03347968
Title: A Phase 1, Open-label Study to Compare the Pharmacokinetics and Pharmacodynamics of Warfarin and Esmolol in the Absence and Presence of MEDI0382 in Healthy Subjects
Brief Title: Study to Compare Pharmacokinetics & Pharmacodynamics of Warfarin & Esmolol in the Absence & Presence of MEDI0382
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5670C00009
Record Dates: First submitted 2017-10-16; First posted 2017-11-20 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteers
Keywords: type 2 Diabetes Mellitus, MEDI0382
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cotadutide; Warfarin; esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MEDI0382 (Experimental): All participants will receive MEDI0382.
  Interventions: Biological: MEDI0382
- Warfarin (Active Comparator): All participants will receive Warfarin
  Interventions: Drug: Warfarin
- Esmolol (Active Comparator): All participants will receive Esmolol
  Interventions: Drug: Esmolol

INTERVENTIONS:
Biological: MEDI0382 — All participants will receive MEDI0382
  Arms: MEDI0382
Drug: Warfarin — All participants will receive Warfarin
  Arms: Warfarin
Drug: Esmolol — All participants will receive Esmolol
  Arms: Esmolol

SUMMARY:
A Phase 1 study to evaluate the effect of MEDI0382 on PK and PD of warfarin and esmolol in healthy subjects.

DETAILED DESCRIPTION:
This is a Phase 1 open label, one-sequence, crossover study to evaluate the effect of MEDI0382 on PK and PD of warfarin and esmolol in healthy subjects. The safety and tolerability of MEDI0382 in combination with warfarin and esmolol will also be evaluated. Following screening, the study consists of 2 5-day inpatient stays followed by outpatient visits.

ELIGIBILITY:
Inclusion Criteria:.

* Healthy volunteers aged ≥ 18 to 45 years
* BMI between 18 -30 kg/m2
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception

Exclusion Criteria:

* Any concurrent condition that in the opinion of the investigator would interfere with the evaluation of the investigational product
* Receipt of investigational product as part of a clinical study or a GLP-1 analogue containing preparation within the last 30 days or 5 half-lives of the drug (whichever is longer) at the time of screening.
* Concurrent participation in another study of any kind
* Severe allergy/hypersensitivity to any of the proposed study treatments or excipients.
* History or presence of gastrointestinal (GI), hepatic, or renal disease or any other conditions known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Impaired renal function is defined as estimated glomerular filtration rate (eGFR) < 60 mL/minute/1.73 m2 at screening.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of screening.
* History of hemophilia, von Willebrand's disease, lupus anticoagulant, or other diseases/syndromes that can either alter or increase the propensity for bleeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Maximum international normalized ratio (INRmax) | Days 2-8 and Days 27-33
  To assess the INR max in the absence and presence of Warfarin on a steady state MEDI0382
Change in heart rate from resting after a 9-minute excercise treadmill test (Bruce Protocol, first 3 stages) | Days 1 and 26
  To assess the effects of MEDI0382 on the hear rate-lowering effect of esmolol during treadmill test.
Maximum international normalized ratio (INRmax) | Days 2-8 and Days 27-33
  To assess the AUC INR in the absence and presence of Warfarin on a steady state MEDI0382

SECONDARY OUTCOMES:
PK(AUC) of R-Warfarin and S-Warfarin | Days 2 and 27
  To assess AUC of R-warfarin and S-warfarin in the presence and absence of steady state MEDI0382
PK (Cmax) of R-Warfarin and S-Warfarin | Days 2 and 27
  To assess Cmax of R-warfarin and S-warfarin in the presence and absence of steady state MEDI0382
Number of patients with Adverse Events (AEs) | 33 Days
  To assess the adverse events as a criteria of safety and tolerability variables.
12 lead electrocardiogram including RR, PR, QRS, QT and QTc intervals | Day 1, Day 8, Day 13, and Day 18
  To assess the cardiovascular system functioning as a criteria of safety and tolerability variables.
Anti-drug antibody titer incidence | Days 1 and 33
  To evaluate the safety and tolerability of multiple doses of MEDI0382 in conjunction with Warfarin and Esmolol.
Clinical laboratory assessments (hematology) | Days 1 and 33
  To assess hematology as a criteria of safety and tolerability variables..
Vital signs (systolic and diastolic blood pressure) | Days 1-8, Days 12 and 13, Days 25-33
  To assess the vital signs as a criteria of safety and tolerability variables
Vital signs (pulse rate and respiratory rate | Days 1-8, Days 12 and 13, Days 25-33
  To assess the vital signs as a criteria of safety and tolerability variables
Clinical laboratory assessments (serum chemistry) | Day -1, Day 8, Day 17, Day 25 and Day 33
  To assess clinical chemistry as a criteria of safety and tolerability variables.
Clinical laboratory assessment (urinalysis) | Day -1
  To assess urinalysis as a criteria of safety and tolerability variables.

CONTACTS AND LOCATIONS:
Overall Officials: Armando Flor, Study Director — MedImmune LLC
Locations (1):
- Research Site, Daytona Beach, Florida, United States